CLINICAL TRIAL: NCT02569710
Title: A Phase 2a, Open-Label Study to Evaluate the Safety, Pharmacokinetics and Efficacy of the Combination of AL-335 and Odalasvir, With or Without Simeprevir, in Treatment-Naïve Subjects With Genotype 1, 2 or 3 Chronic Hepatitis C Infection With or Without Compensated Child Pugh A Cirrhosis
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics and Efficacy of the Combination of AL-335, Odalasvir, and Simeprevir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AL-335-604
Record Dates: First submitted 2015-10-01; First posted 2015-10-07 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — adafosbuvir; odalasvir; Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Cohorts 1 and 2 (Without Cirrhosis) : AL-335+ODV+SMV (Experimental): Treatment-naïve non-cirrhotic Hepatitis C virus (HCV)-infected participants will receive AL-335 and Odalasvir (ODV) with Simeprevir (SMV) for 8 weeks.
  Interventions: Drug: AL-335; Drug: Odalasvir (ODV); Drug: Simeprevir (SMV)
- Cohort 1b (Without Cirrhosis) : AL-335+ODV (Experimental): Treatment-naïve non-cirrhotic HCV-infected participants will receive AL-335 and ODV for 8 weeks.
  Interventions: Drug: AL-335; Drug: Odalasvir (ODV)
- Cohort 3 (Without Cirrhosis) : AL-335+ODV+SMV (Experimental): Treatment-naïve non-cirrhotic HCV-infected participants will receive AL-335 and ODV with SMV for 6 weeks.
  Interventions: Drug: AL-335; Drug: Odalasvir (ODV); Drug: Simeprevir (SMV)
- Cohort 4 (Without Cirrhosis) : AL-335+ODV (Experimental): Treatment-naïve non-cirrhotic HCV-infected participants will receive AL-335 and ODV up to 8 or 12 weeks.
  Interventions: Drug: AL-335; Drug: Odalasvir (ODV)
- Cohort 5 (Without Cirrhosis) : AL-335+ODV + SMV (Experimental): Treatment-naïve non-cirrhotic HCV-infected participants will receive AL-335 and ODV with SMV up to 8 or 12 weeks.
  Interventions: Drug: AL-335; Drug: Odalasvir (ODV); Drug: Simeprevir (SMV)
- Cohorts 6, 7, 8 and 12 (With Cirrhosis) : AL-335+ODV+SMV (Experimental): Treatment naïve or treatment experienced HCV-infected participants with compensated cirrhosis will receive AL-335 and ODV with SMV for 8 weeks.
  Interventions: Drug: AL-335; Drug: Odalasvir (ODV); Drug: Simeprevir (SMV)
- Cohorts 9, 10 and 11 (With Cirrhosis) : AL-335+ODV+SMV (Experimental): Treatment naïve or treatment experienced HCV-infected participants with compensated cirrhosis will receive AL-335 and ODV with SMV for 12 weeks.
  Interventions: Drug: AL-335; Drug: Odalasvir (ODV); Drug: Simeprevir (SMV)
- Cohorts 12 to 15: AL-335+ODV With/without SMV (Experimental): Based on safety, pharmacokinetic (PK), and viral load data, the treatment duration (4 to 12 weeks) and dose levels (AL-335: 400-1,200 milligram [mg], ODV: 25-50 mg with/without SMV: 75-150 mg) may be changed for ongoing and future cohorts (up to 15) after obtaining agreement from the Sponsor and the Principal Investigator.
  Interventions: Drug: AL-335; Drug: Odalasvir (ODV); Drug: Simeprevir (SMV)

INTERVENTIONS:
Drug: AL-335 — AL-335 tablets will be administered in a dose range of 400 to 1200 mg once daily (QD).
Drug: Odalasvir (ODV) — ODV capsules will be administered in a dose range of 25 to 50 mg.
  Other Names: ACH-3102
Drug: Simeprevir (SMV) — SMV tablets will be administered in a dose range of 75 to 150 mg QD or every other day (QOD).
  Arms: Cohort 3 (Without Cirrhosis) : AL-335+ODV+SMV; Cohort 5 (Without Cirrhosis) : AL-335+ODV + SMV; Cohorts 1 and 2 (Without Cirrhosis) : AL-335+ODV+SMV; Cohorts 12 to 15: AL-335+ODV With/without SMV; Cohorts 6, 7, 8 and 12 (With Cirrhosis) : AL-335+ODV+SMV; Cohorts 9, 10 and 11 (With Cirrhosis) : AL-335+ODV+SMV

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of AL-335 in combination with odalasvir (ODV) with or without simeprevir (SMV) in participants with genotype (GT)1 or GT2 or GT3 chronic hepatitis C (CHC) infection.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided written consent
2. In the Investigator's opinion, the participant is able to understand and comply with protocol requirements, instructions, and protocol stated restrictions and is likely to complete the study as planned
3. Male or female, 18-70 years of age
4. Body mass index (BMI) 18-35 kilogram per meter square (kg/m^2), inclusive
5. A woman of childbearing potential must have a negative serum (beta-human chorionic gonadotropin) pregnancy test at screening
6. Female participants must either:

   * not be of childbearing potential defined as: i. Postmenopausal for at least 12 months (that is [i.e.], 2 years of amenorrhea without an alternative medical cause) and a serum follicle stimulating hormone (FSH) level in the postmenopausal range (per reference laboratory), OR ii. Surgically sterile (example [e.g.], underwent total hysterectomy, bilateral oophorectomy, or bilateral tubal ligation/bilateral tubal clips without reversal operation), or otherwise incapable of becoming pregnant, OR
   * be of childbearing potential AND
   * not heterosexually active (e.g., abstinent or homosexual) from screening until 6 months after study drug administration (or longer, if dictated by local regulations), OR
   * if heterosexually active

     * have a vasectomized partner (confirmed sterile per verbal account of the participant), OR
     * using an acceptable method of birth control from screening and agree to continue to use the same method of contraception throughout the study and for 6 months after study drug administration (or longer, if dictated by local regulations). Oral hormone based contraceptives are not allowed from 14 days before the planned study drug administration until 6 months after the last dose of treatment due to the potential for drug-drug interactions which might undermine their efficacy. An intrauterine device (IUD), being either hormonal (i.e., Intra-Uterine System [IUS*]) or non-hormonal, is considered highly effective and reliable; therefore participants using an IUD/IUS are not required to use additional contraceptive methods (no double-barrier method is required). Other non-oral hormone-based contraception methods (e.g., injectable, implants, transdermal system, vaginal ring) may be continued, but as the interaction of the study drug with hormone-based contraception is unknown, these methods are not considered to be reliable and therefore participants should use a double-barrier method (e.g., male condom+either diaphragm or cervical cap with or without spermicide).

       * An IUS does not rely on systemic plasma concentrations and is therefore not expected to be impacted by a potential drug-drug interaction (DDI)

   Note 1: Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.

   Note 2: A male and female condom should not be used together due to risk of breakage or damage caused by latex friction
7. A post-menopausal female who is receiving hormone replacement therapy and is willing to discontinue hormone therapy 30 days before study drug dosing and agrees to remain off hormone replacement therapy for the duration of the study may be eligible for study participation.

   * Male participants must either:
   * be surgically sterile (had a vasectomy), or otherwise incapable of fathering a child, OR
   * not be heterosexually active (e.g., abstinent or homosexual) from enrollment (Day 1) in the study until at least 6 months after study drug administration, OR
   * if heterosexually active:

     * have a partner who is postmenopausal (2 years amenorrhea), surgically sterile (e.g., has had a total hysterectomy, bilateral oophorectomy, or bilateral tubal ligation/bilateral tubal clips without reversal operation), or otherwise incapable of becoming pregnant OR
     * be practicing an acceptable method of birth control from enrollment in the study (Day 1) and agree to continue to use the same method of contraception throughout the study and for at least 6 months after study drug administration (or longer, if dictated by local regulations). An acceptable method of birth control for male participants is a double-barrier method (e.g., male condom+either diaphragm or cervical cap with or without spermicide).

   Note: Male participants with a female partner who uses hormonal contraceptives (oral, injectable, implants) or a hormonal (IUS) or non-hormonal IUD and male participants who are vasectomized or otherwise incapable of fathering a child are not required to use additional contraceptive methods.

   Note 1: Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.

   Note 2: A male and female condom should not be used together due to risk of breakage or damage caused by latex friction.

   NOTE: Contraceptive use by men and women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies if these are stricter than what is proposed in these inclusion criteria
8. Participants must agree to refrain from sperm/egg donation from start of dosing through 6 months after the completion of study drug administration
9. Genotype (GT) 1a or 1b or GT2 or 3 chronic hepatitis C (CHC), depending on cohort, with positive Hepatitis C virus (HCV) antibody and a positive HCV ribonucleic acid (RNA) at screening including documentation of CHC infection for at least 6 months. Genotype testing must occur at a screening visit. NOTE: GT1 patients are eligible for inclusion even if they cannot be successfully subtyped unless a specific subtype is required for a cohort
10. Screening HCV RNA viral load greater than or equal to (>=) 50,000 International Units per milliliter (IU/mL), except for participants with compensated cirrhosis (Child Pugh Class A) who may have HCV RNA viral load >=10^4 IU/mL
11. No prior treatment for CHC (defined as no prior exposure to any approved or investigational drug including direct-acting antivirals, and interferon-based treatments)
12. Fibroscan, collected within 6 months of baseline visit, with liver stiffness score less than or equal to (<=) 12.5 kilo Pascal (kPa) to be eligible (except for participants with cirrhosis, see below).

    * participants with compensated cirrhosis must meet the Child-Pugh Class A definition (see Appendix G) and at least one of the following criteria: i. Liver biopsy result indicating the presence of cirrhosis (e.g., Metavir F4; Ishak >5) or ii. Fibroscan evaluation with a liver stiffness score >12.5 kPa
13. Participant is otherwise in good health as deemed by the investigator, based on the findings of a medical evaluation including medical history, physical examination, laboratory tests and electrocardiogram (ECG)
14. Willing to avoid prolonged sun exposure and use of tanning devices while taking Simeprevir (SMV) and through 4 weeks of follow up. Participant should also be advised to use a broad-spectrum sunscreen and lip balm of at least sun protection factor >30 to help protect against potential sunburn

Exclusion Criteria:

1. Pregnant, planning on becoming pregnant (during treatment and up to 6 months after the end of treatment [EOT]), or breast-feeding female participant, or male participant whose female partner is pregnant or planning on becoming pregnant (during treatment and up to 6 months after the EOT)
2. Other than CHC with or without compensated cirrhosis, clinically significant cardiovascular, respiratory, renal, gastrointestinal, hematologic, neurologic, thyroid or any other medical illness or psychiatric disorder, as determined by the Investigator and/or Sponsor's Medical Monitor
3. History or other clinical evidence of significant or unstable cardiac disease (e.g., angina, congestive heart failure, myocardial infarction, diastolic dysfunction, significant arrhythmia, coronary heart disease, and/or clinically significant ECG abnormalities), moderate to severe valvular disease or uncontrolled hypertension at screening
4. Screening echocardiogram ejection fraction <55 percentage (%) or any other echocardiographic finding suggestive of clinically relevant cardiomyopathy
5. Creatinine clearance of <60 mL/min (Cockcroft-Gault)
6. Positive test for Hepatitis A virus immunoglobulin (HAV) Immunoglobulin M (IgM), Hepatitis B surface antigen (HBsAg), or Human Immunodeficiency Virus (HIV) Ab
7. Abnormal screening laboratory results that are considered clinically significant by the investigator
8. History of clinical hepatic decompensation, e.g., variceal bleeding, spontaneous bacterial peritonitis, ascites, hepatic encephalopathy or active jaundice (within last year)
9. Any condition that, in the opinion of the investigator, would compromise the study's objectives or the well-being of the participant or prevent the participant from meeting the study requirements
10. Participation in an investigational drug trial or having received an investigational vaccine within 30 days or 5 half lives (whichever is longer) prior to study medication
11. Clinically significant abnormal screening ECG findings (e.g., PR >200 msec, QRS interval >120 millisecond (msec) or corrected QT interval (QTc) >450 msec for male participants and >470 msec for female participants), based on an average of triplicate ECGs. Any evidence of heart block or bundle branch block is also exclusionary
12. History or family history of abnormal ECG intervals, for example prolonged QT syndrome (torsade de pointes) or sudden cardiac death
13. The participant has a positive prestudy drug screen, including methadone unless the drug is prescribed by the participant's physician. The list of drugs that should be screened for includes amphetamines, barbiturates, cocaine, opiates, phencyclidine (PCP), and benzodiazepines
14. Laboratory abnormalities including:

    * Hematocrit <0.34
    * White blood cell counts <3,500/millimeter (mm)^3 (<1,000/mm^3 for participants with compensated cirrhosis)
    * Absolute neutrophil count <1,000/mm^3 (<750/mm^3 for participants with compensated cirrhosis)
    * Platelets <=120,000/mm^3 (platelets ≤90,000/mm^3 for participants with compensated cirrhosis)
    * Glycosylated hemoglobin (HbA1C) >55 mmol/mol
    * Prothrombin time >=1.5 * upper limit of normal (ULN)
    * Albumin <=32 gram per liter (g/L), bilirubin >=1.5 milligram per deciliter (mg/dL) at screening (participants with documented Gilbert's disease allowed)
    * Serum ALT concentration >=5* ULN
    * CK >1.5* ULN A single repeat laboratory evaluation under appropriate conditions (e.g., fasted, no antecedent exercise) is allowed for eligibility determination
15. Any condition possibly affecting drug absorption (e.g., gastrectomy or other significant gastrointestinal tract surgery, such as gastroenterostomy, small bowel resection, or active enterostomy)
16. Clinically significant blood loss or elective blood donation of significant volume (i.e., >500 mL) within 60 days of first dose of study drug; >1 unit of plasma within 7 days of first dose of study drug
17. Evidence of clinically relevant active infection that would interfere with study conduct or its interpretation
18. History of regular alcohol intake >10 standard drinks per week of alcohol for females and >15 standard drinks per week for males (one unit is defined as 10 g alcohol) within 3 months of the screening visit
19. The use of prohibited medications, including prescription, over the counter (OTC) medications, herbal medications, inducers or inhibitors of Cytochrome P450 (CYP450) enzymes or drug transporters (including P-gp) within 14 days prior to the first dose of study medication is excluded, unless previously approved by the Sponsor's Medical Monitor. NOTE: Chronic medication use is permitted so long as they are medically necessary, deemed acceptable by the Principal Investigator and Medical Monitor, and not Prohibited Medications (see Section 5.12)
20. Hypersensitivity to the active substances (including sulfa allergy) or to any of the excipients of AL-335, Odalasvir (ODV) or SMV
21. Evidence on recent (within 6 months) liver ultrasound of hepatic mass or lesion concerning for malignancy (participants with cirrhosis only)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2015-10-31 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alios Biopharma Inc. Clinical Trial, Study Director — Alios Biopharma Inc.
Locations (11):
- CAP Research Ltd, Phoenix, Mauritius
- Republican Clinical Hospital, Chisinau, Moldova
- New Zealand (6):
  - Auckland Clinical Studies, Auckland
  - Christchurch Clinical Studies Trust, Christchurch
  - Waikato Hospital, Hamilton
  - P3 Research Ltd - Hawkes Bay, Havelock North
  - P3 Research Ltd - Wellington, Wellington
  - Wellington Hospital, Wellington
- United Kingdom (3):
  - King's College Hospital, Brixton
  - NHS Greater Glasgow and Clyde Glasgow Royal Infirmary, Glasgow
  - Pennine Acute Hospitals Trust, Oldham

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No participants were recruited for Cohorts 10 and 12, hence no data is reported here for these two cohorts.
Groups:
- Cohort 1 (8 Weeks Genotype [GT1]): Cohort 1 (Participants without Cirrhosis) received single dose of AL-335 400 milligrams (mg) tablets once daily (QD), odalasvir (ODV) 50 mg tablet and simeprevir 100 mg tablet QD for 8 weeks.
- Cohort 1b + Cohort 4 (8 Weeks GT1): Cohort 1b (Participants without Cirrhosis) received single dose of AL-335 800 mg tablets QD and ODV 50 mg tablets every other day (QOD) for 8 weeks; Cohort 4 (Participants without Cirrhosis) received single dose of AL-335 800 mg tablets QD and ODV 50 mg tablets QOD for 8 weeks.
- Cohort 2 (8 Weeks GT1): Cohort 2 (Participants without Cirrhosis) received single dose of AL-335 800 mg tablets QD, ODV 50 mg tablets QOD and SMV 75 mg tablets QD for 8 weeks.
- Cohort 3 (6 Weeks GT1): Cohort 3 (Participants without Cirrhosis) received single dose of AL-335 800 mg QD, ODV 50 mg QOD and SMV 75 mg QD for 6 weeks.
- Cohort 4 (12 Weeks GT1): Cohort 4 (Participants without Cirrhosis) received single dose of AL-335 800 mg tablets QD and ODV 50 mg tablets QOD for 12 weeks.
- Cohort 5a (8 Weeks GT3): Cohort 5 (Participants without Cirrhosis) received single dose of AL-335 800 mg tablets QD, ODV 50 mg tablets QOD and SMV 75 mg tablets QD for 8 weeks.
- Cohort 5b (12 Weeks GT3): Cohort 5 (Participants without Cirrhosis) received single dose of AL-335 800 mg tablets QD, ODV 50 mg tablets QOD and SMV 75 mg tablets QD for 12 weeks.
- Cohort 6,7,8 (8 Weeks GT1 F4): Cohort 6 (Participants with Cirrhosis) received single dose of AL-335 800 mg tablets QD, ODV 50 mg tablets QOD and SMV 75 mg tablets QD for 8 weeks; Cohort 7 and Cohort 8 (Participants with Cirrhosis) received single dose of AL-335 800 mg tablets QD, ODV 25 mg tablets QD and SMV 75 mg tablets QD for 8 weeks.
- Cohort 9 (12 Weeks GT1 F4): Cohort 9 (Participants with Cirrhosis) received single dose of AL-335 800 mg tablets QD, ODV 25 mg tablets QD and SMV 75 mg tablets QD for 12 weeks.
- Cohort 11 (12 Weeks GT2 F4): Cohort 11 (Participants with Cirrhosis) received single dose of AL-335 800 mg tablets QD, ODV 25 mg tablets QD and SMV 75 mg tablets QD for 12 weeks.
Period: Overall Study
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Started | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Completed | 19 | 25 | 20 | 20 | 7 | 4 | 12 | 30 | 14 | 4
Not Completed | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Virologic failure | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4) | Total
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4 | 161
Age, Continuous [Median (Full Range); unit: years] | 56 [30 to 61] | 55 [29 to 64] | 56 [36 to 62] | 55.5 [30 to 64] | 55 [41 to 60] | 54 [38 to 64] | 44.5 [18 to 65] | 56.5 [37 to 68] | 52 [36 to 67] | 63.5 [61 to 69] | 55 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 6 | 8 | 5 | 0 | 1 | 16 | 2 | 1 | 54
  Male | 13 | 17 | 14 | 12 | 3 | 5 | 13 | 14 | 13 | 3 | 107
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 17 | 18 | 14 | 6 | 2 | 12 | 27 | 9 | 3 | 128
  Asian | 0 | 4 | 1 | 2 | 0 | 2 | 1 | 1 | 1 | 1 | 13
  Native Hawaiian or other Pacific Islander | 0 | 3 | 0 | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 10
  Multiple | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Other | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 5 | 0 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Moldova | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 3 | 0 | 16
  Mauritius | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 0 | 8
  New Zealand | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 14 | 5 | 3 | 134

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Event (TEAE)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent were events between administration of study drug and up to 43 weeks that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Up to 43 weeks
Population: Safety set included all participants enrolled into the study who had received at least 1 dose of any study drug, whether prematurely withdrawn from the study or not.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Participants | 17 | 19 | 14 | 13 | 7 | 4 | 13 | 17 | 10 | 4

2. Primary Outcome: Body Weight at End of Treatment
Description: Body weight (measured using a calibrated scale) at end of treatment was reported.
Time Frame: End of treatment (Cohort 3: 6 weeks; Cohort 1, Cohort 1b+ Cohort 4, Cohort 2, Cohort 5a, and Cohort 6, 7, 8: 8 weeks; Cohort 4, Cohort 5b, Cohort 9 and Cohort 11: 12 weeks)
Population: Safety set included all participants enrolled into the study who had received at least 1 dose of any study drug, whether prematurely withdrawn from the study or not. Here, N (number of participants analyzed) signifies number of participants evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 19 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Kilograms (kg) | 76.02 (15.13) | 84.58 (15.09) | 80.19 (17.79) | 74.07 (12.78) | 73.09 (8.62) | 81.30 (13.82) | 81.83 (13.67) | 80.15 (17.92) | 86.02 (15.56) | 69.90 (11.55)

3. Primary Outcome: Body Mass Index (BMI) at End of Treatment
Description: BMI was calculated by dividing the body weight (in kilogram) by the square of height (in meters). BMI at end of treatment was reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms per square meter (Kg/m^2)
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 19 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Kilograms per square meter (Kg/m^2) | 25.89 (4.63) | 28.43 (4.26) | 26.45 (5.53) | 25.46 (3.53) | 25.60 (3.21) | 25.60 (2.82) | 26.17 (4.20) | 27.69 (5.28) | 27.98 (4.37) | 23.64 (4.50)

4. Primary Outcome: Percentage of Participants With Worst Post-Baseline Values of Vital Signs
Description: Percentage of participants with worst post-baseline values of vital signs (Systolic blood pressure [sBP], Diastolic blood pressure [dBP], and Heart rate) were reported. For sBP, abnormally low: less than or equal to [<=] 90 millimeters mercury [mmHg]; Grade 1 or mild: greater than [>] 140 to less than [<] 160 mmHg; Grade 2 or moderate: >=160 to <180 and Grade 3 or severe: >=180 mmHg. For dBP, abnormally low: <=50 mmHg; Grade 1 or mild: >90 to <100 mmHg; Grade 2 or moderate: >=100 to <110 mmHg and Grade 3 or severe: >=110 mmHg. For Heart Rate, abnormally low: <=50 beats per minute [bpm] and abnormally high: >=120 bpm.
Time Frame: Up to 43 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Percentage of participants
  sBP: Abnormally low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3.3 | 0 | 0
  sBP: Grade 1 or mild | 20.0 | 32.0 | 35.0 | 25.0 | 37.5 | 60.0 | 57.1 | 26.7 | 46.7 | 25.0
  sBP: Grade 2 or moderate | 10.0 | 8.0 | 0 | 5.0 | 37.5 | 0 | 7.1 | 20.0 | 13.3 | 50.0
  sBP: Grade 3 or severe | 0 | 4.0 | 5.0 | 0 | 0 | 0 | 0 | 3.3 | 13.3 | 0
  dBP: Abnormally low | 0 | 4.0 | 0 | 0 | 12.5 | 0 | 0 | 0 | 0 | 0
  dBP: Grade 1 or mild | 5.0 | 20.0 | 35.0 | 20.0 | 0 | 60.0 | 21.4 | 10.0 | 26.7 | 0
  dBP: Grade 2 or moderate | 5.0 | 12.0 | 0 | 0 | 0 | 0 | 14.3 | 13.3 | 6.7 | 25.0
  dBP: Grade 3 or severe | 0 | 0 | 0 | 0 | 25.0 | 0 | 7.1 | 3.3 | 6.7 | 0
  Heart Rate: Abnormally low | 35.0 | 32.0 | 35.0 | 30.0 | 50.0 | 20.0 | 21.4 | 13.3 | 13.3 | 0
  Heart Rate: Abnormally high | 0 | 0 | 0 | 0 | 12.5 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Percentage of Participants With Maximum Decrease From Baseline in Mean Ejection Fraction
Description: Percentage of participants with maximum decrease from baseline in mean ejection fraction was reported. Percentages are based on the number of participants with available data.
Time Frame: Baseline up to End of treatment (up to 43 weeks)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Percentage of participants
  Decline of > 10% | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Decline of >5-<=10% | 0.0 | 4.0 | 10.0 | 10.0 | 12.5 | 0.0 | 21.4 | 3.3 | 6.7 | 0.0
  Decline of >0-<=5% | 65.0 | 48.0 | 60.0 | 50.0 | 50.0 | 20.0 | 64.3 | 80.0 | 46.7 | 50.0

6. Primary Outcome: Percentage of Participants by Treatment Emergent Toxicity Grade - Hematology Parameters
Description: Percentage of participants by treatment emergent toxicity grade (1, 2, 3, 4 and 3+4) for Hematology parameters (hemoglobin, lymphocytes, neutrophils, leukocytes, platelets) were reported. Toxicity grades were defined as Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe and Grade 4: potentially life-threatening. A toxicity is treatment-emergent if it is worse than the baseline or if baseline is missing.
Time Frame: Up to 43 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Percentage of participants
  Hemoglobin: Grade 1 | 5.0 | 0.0 | 0.0 | 5.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Hemoglobin: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Hemoglobin: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Hemoglobin: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Hemoglobin: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Lymphocytes: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.7 | 0.0 | 0.0
  Lymphocytes: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 7.1 | 10.0 | 0.0 | 0.0
  Lymphocytes: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Lymphocytes: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Lymphocytes: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Neutrophils: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0
  Neutrophils: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Neutrophils: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Neutrophils: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Neutrophils: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Leukocytes: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 10.0 | 0.0 | 0.0
  Leukocytes: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Leukocytes: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Leukocytes: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Leukocytes: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Platelets: Grade 1 | 5.0 | 0.0 | 5.0 | 5.0 | 0.0 | 0.0 | 7.1 | 6.7 | 13.3 | 25.0
  Platelets: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 16.7 | 0.0 | 0.0
  Platelets: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Platelets: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Platelets: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

7. Primary Outcome: Percentage of Participants by Treatment Emergent Toxicity Grade - Blood Chemistry Parameters
Description: Percentage of participants by treatment emergent toxicity grade (Grade 1,2,3,4,3+4) for Blood Chemistry (Calcium, Phosphate, Potassium, Sodium, Bicarbonate, Alanine aminotransferase, Alkaline phosphatase, Aspartate aminotransferase, Bilirubin, Direct bilirubin, Glucose, Cholesterol, Triglycerides, Urate, Triacylglycerol lipase, Creatinine, Creatinine clearance, Albumin and Creatine kinase) were reported. Toxicity grades were defined as Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe and Grade 4: potentially life-threatening. A toxicity is treatment-emergent if it is worse than the baseline or if baseline is missing.
Time Frame: Up to 43 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Percentage of participants
  Calcium: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 13.3 | 0.0 | 0.0
  Calcium: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Calcium: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Calcium: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Calcium: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Phosphate: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Phosphate: Grade 2 | 10.0 | 20.0 | 25.0 | 15.0 | 12.5 | 0.0 | 14.3 | 13.3 | 6.7 | 0.0
  Phosphate: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 21.4 | 3.3 | 0.0 | 0.0
  Phosphate: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Phosphate: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 21.4 | 3.3 | 0.0 | 0.0
  Potassium: Grade 1 | 0.0 | 4.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.7 | 0.0 | 0.0
  Potassium: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Potassium: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Potassium: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Potassium: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Sodium: Grade 1 | 0.0 | 8.0 | 5.0 | 0.0 | 12.5 | 20.0 | 0.0 | 3.3 | 20.0 | 0.0
  Sodium: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Sodium: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Sodium: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Sodium: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Bicarbonate: Grade 1 | 0.0 | 16.0 | 15.0 | 5.0 | 12.5 | 20.0 | 7.1 | 0.0 | 0.0 | 0.0
  Bicarbonate: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.7 | 0.0 | 0.0
  Bicarbonate: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Bicarbonate: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Bicarbonate: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Alanine aminotransferase: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0
  Alanine aminotransferase: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Alanine aminotransferase: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Alanine aminotransferase: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.7 | 0.0 | 0.0
  Alanine aminotransferase: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.7 | 0.0 | 0.0
  Alkaline phosphatase: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.7 | 0.0 | 0.0
  Alkaline phosphatase: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Alkaline phosphatase: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Alkaline phosphatase: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Alkaline phosphatase: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Aspartate aminotransferase: Grade: 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 25.0
  Aspartate aminotransferase: Grade: 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0
  Aspartate aminotransferase: Grade: 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.7 | 0.0
  Aspartate aminotransferase: Grade: 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Aspartate aminotransferase: Grade: 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.7 | 0.0
  Bilirubin: Grade 1 | 0.0 | 0.0 | 10.0 | 10.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0
  Bilirubin: Grade 2 | 5.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 25.0
  Bilirubin: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0
  Bilirubin: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Bilirubin: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0
  Direct bilirubin: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Direct bilirubin: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Direct bilirubin: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 6.7 | 0.0
  Direct bilirubin: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Direct bilirubin: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 6.7 | 0.0
  Glucose: Grade 1 | 15.0 | 4.0 | 10.0 | 5.0 | 25.0 | 0.0 | 35.7 | 10.0 | 13.3 | 0.0
  Glucose: Grade 2 | 0.0 | 4.0 | 5.0 | 0.0 | 12.5 | 0.0 | 14.3 | 13.3 | 13.3 | 25.0
  Glucose: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0
  Glucose: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Glucose: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0
  Cholesterol: Grade 1 | 20.0 | 24.0 | 30.0 | 35.0 | 12.5 | 0.0 | 42.9 | 3.3 | 20.0 | 50.0
  Cholesterol: Grade 2 | 15.0 | 8.0 | 5.0 | 5.0 | 37.5 | 0.0 | 0.0 | 6.7 | 6.7 | 0.0
  Cholesterol: Grade 3 | 0.0 | 0.0 | 5.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0
  Cholesterol: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Cholesterol: Grade 3+4 | 0.0 | 0.0 | 5.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0
  Triglycerides: Grade 1 | 5.0 | 16.0 | 10.0 | 15.0 | 50.0 | 20.0 | 28.6 | 16.7 | 33.3 | 25.0
  Triglycerides: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 14.3 | 0.0 | 0.0 | 0.0
  Triglycerides: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Triglycerides: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Triglycerides: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Urate: Grade 1 | 5.0 | 12.0 | 5.0 | 0.0 | 12.5 | 0.0 | 28.6 | 10.0 | 26.7 | 0.0
  Urate: Grade 2 | 0.0 | 4.0 | 0.0 | 5.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0
  Urate: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Urate: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Urate: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Triacylglycerol lipase: Grade 1 | 5.0 | 12.0 | 5.0 | 0.0 | 12.5 | 20.0 | 7.1 | 13.3 | 0.0 | 0.0
  Triacylglycerol lipase: Grade 2 | 15.0 | 4.0 | 10.0 | 0.0 | 12.5 | 0.0 | 7.1 | 3.3 | 0.0 | 0.0
  Triacylglycerol lipase: Grade 3 | 5.0 | 8.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Triacylglycerol lipase: Grade 4 | 0.0 | 0.0 | 5.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Triacylglycerol lipase: Grade 3+4 | 5.0 | 8.0 | 5.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Creatinine: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Creatinine: Grade 2 | 0.0 | 0.0 | 0.0 | 5.0 | 0.0 | 0.0 | 7.1 | 0.0 | 0.0 | 0.0
  Creatinine: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 12.5 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0
  Creatinine: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Creatinine: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 12.5 | 0.0 | 0.0 | 3.3 | 0.0 | 0.0
  Creatinine clearance: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Creatinine clearance: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 20.0 | 0.0
  Creatinine clearance: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Creatinine clearance: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Creatinine clearance: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Albumin: Grade 1 | 5.0 | 4.0 | 0.0 | 0.0 | 25.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Albumin: Grade 2 | 0.0 | 8.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Albumin: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Albumin: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Albumin: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Creatine kinase: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 7.1 | 0.0 | 0.0 | 0.0
  Creatine kinase: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.7 | 0.0
  Creatine kinase: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Creatine kinase: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Creatine kinase: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

8. Primary Outcome: Percentage of Participants by Treatment Emergent Toxicity Grade - Prothrombin International Normalized Ratio (INR)
Description: Percentage of participants by treatment emergent toxicity grade for coagulation parameter (Prothrombin International Normalized Ratio) were reported. Toxicity grades were defined as Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe and Grade 4: potentially life-threatening. A toxicity is treatment-emergent if it is worse than the baseline or if baseline is missing.
Time Frame: Up to 43 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Percentage of participants
  Prothrombin INR: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Prothrombin INR: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Prothrombin INR: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Prothrombin INR: Grade 4 | 0.0 | 4.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Prothrombin INR: Grade 3+4 | 0.0 | 4.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

9. Primary Outcome: Percentage of Participants by Treatment Emergent Toxicity Grade - Urinalysis Parameter (Protein)
Description: Percentage of participants by treatment emergent toxicity grade (Grade 1, 2, 3, 4, 3+4) for urinalysis parameter (protein) was reported. Toxicity grades were defined as Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe and Grade 4: potentially life-threatening. A toxicity is treatment-emergent if it is worse than the baseline or if baseline is missing.
Time Frame: Up to 43 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Percentage of participants
  Protein: Grade 1 | 0.0 | 4.0 | 0.0 | 0.0 | 0.0 | 0.0 | 7.1 | 3.3 | 26.7 | 50.0
  Protein: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 13.3 | 0.0
  Protein: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 25.0
  Protein: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Protein: Grade 3+4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.3 | 0.0 | 25.0

10. Primary Outcome: Percentage of Participants With Worst Treatment Emergent Abnormalities of Electrocardiogram (ECG) Parameters
Description: Percentage of participants with worst treatment emergent abnormalities of ECG parameters (Fridericia Corrected QT interval [QTcF], Bazett Corrected QT interval [QTcB], Heart rate, QRS and PR, was reported. For QTcF abnormality was defined as 30 milliseconds (ms) less than or equal to (<=) QTcF increase from baseline <= 60 ms; for QTcB abnormality was defined as 30 ms <= QTcB increase from baseline <= 60 ms; for heart rate - abnormal low: <= 50 beats per minute (bpm) and abnormal high: >= 120 bpm; for QRS - abnormal high: >120 ms; for PR - abnormally low: PR < 120 ms; abnormally high - 200 ms < PR <= 240 ms and 240 ms < PR <= 300 ms.
Time Frame: Up to 43 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Percentage of participants
  QTcF: Abnormal | 5.0 | 0.0 | 5.0 | 0.0 | 0.0 | 0.0 | 7.1 | 3.3 | 0.0 | 0.0
  QTcB: Abnormal | 5.0 | 8.0 | 10.0 | 0.0 | 0.0 | 0.0 | 28.6 | 3.3 | 6.7 | 0.0
  Heart rate: Abnormal low | 25.0 | 16.0 | 10.0 | 15.0 | 25.0 | 20.0 | 14.3 | 13.3 | 0.0 | 25.0
  Heart rate: Abnormal high | 0.0 | 0.0 | 0.0 | 0.0 | 12.5 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  QRS: Abnormal high | 0.0 | 4.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  PR: Abnormally low (PR<120 ms) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 7.1 | 3.3 | 0.0 | 0.0
  PR: Abnormally high (200 ms<PR<= 240 ms) | 5.0 | 8.0 | 15.0 | 10.0 | 0.0 | 0.0 | 0.0 | 6.7 | 13.3 | 0.0
  PR: Abnormal high (240 ms<PR<=300 ms) | 10.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 7.1 | 0.0 | 0.0 | 0.0

11. Secondary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at Week 4, 12 and 24 After End of Treatment
Description: Participants were considered to have achieved SVR if the Hepatitis C virus (HCV) Ribonucleic acid (RNA) less than (<) Lower limit of quantification (LLOQ) (<15 international unit per milliliter [IU/mL]) detectable or undetectable at Week 4, 12 and 24 after the actual end of study drug treatment.
Time Frame: At Week 4, 12 and Week 24 after end of treatment (Cohort 3: 6 weeks; Cohort 1, Cohort 1b+ Cohort 4, Cohort 2, Cohort 5a, and Cohort 6, 7, 8: 8 weeks; Cohort 4, Cohort 5b, Cohort 9 and Cohort 11: 12 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Percentage of participants
  4 weeks after end of treatment | 100 [83.2 to 100] | 96.0 [79.6 to 99.9] | 100 [83.2 to 100] | 100 [83.2 to 100] | 87.5 [47.3 to 99.7] | 0 [NA to NA] — NA indicates that upper and lower limit of confidence interval (CI) was not estimable as no participant achieved SVR in this group. | 71.4 [41.9 to 91.6] | 100 [88.4 to 100] | 93.3 [68.1 to 99.8] | 100 [39.8 to 100]
  12 weeks after end of treatment | 100 [83.2 to 100] | 84.0 [63.9 to 95.5] | 100 [83.2 to 100] | 100 [83.2 to 100] | 87.5 [47.3 to 99.7] | 0 [NA to NA] — NA indicates that upper and lower limit of CI was not estimable as no participant achieved SVR in this group. | 71.4 [41.9 to 91.6] | 96.7 [82.8 to 99.9] | 93.3 [68.1 to 99.8] | 100 [39.8 to 100]
  24 weeks after end of treatment | 100 [83.2 to 100] | 84.0 [63.9 to 95.5] | 100 [83.2 to 100] | 100 [83.2 to 100] | 87.5 [47.3 to 99.7] | 0 [NA to NA] — NA indicates that upper and lower limit of CI was not estimable as no participant achieved SVR in this group. | 71.4 [41.9 to 91.6] | 96.7 [82.3 to 99.9] | 93.3 [68.1 to 99.8] | 100 [39.8 to 100]

12. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of AL-335 and Its Metabolites (ALS-022399 and ALS-022227)
Description: Cmin is the minimum observed plasma concentration of AL-335 and its metabolites (ALS-022399 and ALS-022227). For Pharmacokinetic (PK) analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, and 24 hours postdose (Week 2), 2-4 hours postdose (Weeks 3 and 6), 6-8 hours postdose (Weeks 4 and 8)
Population: PK set: all safety set participants except those who violated inclusion/exclusion criteria, deviated from protocol, or if data were unavailable/incomplete which influenced PK analysis.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/ml)
Groups:
- Cohort 1: Cohort 1 (Participants without Cirrhosis) received single dose of AL-335 400 milligrams (mg) tablets once daily (QD), odalasvir (ODV) 50 mg tablet and simeprevir 100 mg tablet QD for 8 weeks.
- Cohort 1b + Cohort 4: Cohort 1b (Participants without Cirrhosis) received single dose of AL-335 800 mg tablets QD and ODV 50 mg tablets every other day (QOD) for 8 weeks; Cohort 4 (Participants without Cirrhosis) received single dose of AL-335 800 mg tablets QD and ODV 50 mg tablets QOD for 8 weeks.
- Cohort 2 + Cohort 3 + Cohort 5: Cohort 2+3+5 (Participants with Cirrhosis): Participants received single dose of AL-335 800 mg QD, ODV 50 mg QOD and SMV 75 mg QD.
- Cohort 6: Cohort 6 (Participants with Cirrhosis) received single dose of AL-335 800 mg QD, ODV 50 mg QOD and SMV 75 mg QD for 8 weeks.
- Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11: Cohort 7+8+9+11 (Participants with Cirrhosis): Participants received single dose of AL-335 800 mg QD, ODV 25 mg QD and SMV 75 mg QD.
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
nanogram per milliliter (ng/ml)
  AL-335 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  ALS-022399 | 0.000 (0.000) | 0.000 (0.000) | 0.308 (1.233) | 0.000 (0.000) | 0.280 (0.814)
  ALS-022227 | 35.73 (13.61) | 35.80 (11.15) | 57.25 (31.63) | 68.30 (38.33) | 64.96 (28.63)

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of AL-335 and Its Metabolites (ALS-022399 and ALS-022227)
Description: Cmax is the maximum observed plasma concentration of AL-335 and its metabolites (ALS-022227). For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
ng/mL
  AL-335 | 414.79 (317.93) | 547.36 (226.06) | 563.04 (423.53) | 529.17 (265.17) | 677.59 (554.83)
  ALS-022399 | 103.57 (52.25) | 148.89 (48.77) | 174.89 (87.05) | 158.80 (55.97) | 186.28 (113.18)
  ALS-022227 | 364.4 (129.1) | 392.6 (144.2) | 658.0 (275.1) | 643.2 (318.4) | 619.7 (224.1)

14. Secondary Outcome: Trough Plasma Concentration (Ctrough) for AL-335 and Its Metabolites (ALS-022399 and ALS-022227)
Description: Ctrough is the trough plasma concentration for AL-335 and its metabolites (ALS-022399 and ALS-022227). For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: PK set: all safety set participants except those who violated inclusion/exclusion criteria, deviated from protocol, or if data were unavailable/incomplete which influenced PK analysis. Here, 'n' signifies the number of participants analyzed for specified analyte.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
ng/ml
  AL-335: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  ALS-022399: number analyzed (Participants) | 0 | 0 | 6 | 2 | 8
  ALS-022399 |  |  | 4.640 (4.018) | 4.570 (2.899) | 4.400 (2.560)
  ALS-022227 | 42.74 (19.26) | 36.77 (10.42) | 61.82 (35.47) | 86.20 (56.31) | 73.85 (35.15)

15. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of AL-335 and Its Metabolites (ALS-022399 and ALS-022227)
Description: Tmax is the time to reach the maximum plasma concentration of AL-335, ALS-022399 and ALS-022227. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (Full Range); unit: Hours
Groups:
- Cohort 2 + Cohort 3 + Cohort 5: Cohort 2+3+5 (Participants without Cirrhosis): Participants received single dose of AL-335 800 mg QD, ODV 50 mg QOD and SMV 75 mg QD
- Cohort 6: Cohort 6 (Participants with Cirrhosis): received single dose of AL-335 800 mg QD, ODV 50 mg QOD and SMV 75 mg QD for 8 weeks.
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
Hours
  AL-335 | 2.000 [0.50 to 4.00] | 2.000 [1.00 to 4.00] | 1.500 [1.00 to 4.00] | 1.000 [1.00 to 2.00] | 2.000 [0.50 to 4.00]
  ALS-022399 | 3.0 [1.00 to 6.00] | 3.000 [2.00 to 4.00] | 3.000 [1.00 to 4.00] | 2.000 [1.00 to 4.00] | 3.000 [2.00 to 6.00]
  ALS-022227 | 4.000 [2.00 to 4.60] | 4.000 [3.00 to 6.00] | 3.500 [2.00 to 6.00] | 3.500 [2.00 to 6.00] | 4.000 [2.00 to 6.00]

16. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Last Measurable Plasma Concentration (AUC [0-last]) of AL-335 and Its Metabolites (ALS-022399 and ALS-022227)
Description: AUC(0-last) is the area under the plasma concentration-time curve from time 0 to last measurable plasma concentration of AL-335, ALS-022399 and ALS-022227. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanogram*hours per milliliters (ng*h/mL)
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
nanogram*hours per milliliters (ng*h/mL)
  AL-335 | 1049.3 (890.0) | 1185.8 (502.8) | 1526.3 (1328.9) | 1178.5 (594.0) | 1774.8 (1348.5)
  ALS-022399 | 469.3 (224.0) | 660.7 (211.5) | 945.2 (551.1) | 844.2 (287.9) | 933.3 (544.3)
  ALS-022227 | 2920.0 (1029.1) | 3238.2 (972.8) | 5258.1 (1969.4) | 5218.3 (2011.9) | 5425.2 (1878.2)

17. Secondary Outcome: Area Under the Plasma Concentration Time-Curve at 24 Hours (AUC0-24) for AL-335 and Its Metabolites (ALS-022399 and ALS-022227)
Description: AUC(0-24) is the area under the plasma concentration-time curve from time zero to time 24 hours for AL-335, ALS-022399 and ALS-022227. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, and 24 hours postdose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
ng*h/mL
  AL-335 | 1058.0 (886.9) | 1197.2 (507.7) | 1532.7 (1329.5) | 1187.3 (600.9) | 1792.2 (1350.9)
  ALS-022399 | 500.5 (230.8) | 718.0 (240.7) | 1009.7 (599.4) | 932.7 (330.1) | 1044.7 (561.1)
  ALS-022227 | 2897.0 (1081.8) | 3238.2 (972.8) | 5258.1 (1969.4) | 4806.0 (1945.4) | 5425.2 (1878.2)

18. Secondary Outcome: Last Measurable Plasma Concentration (Clast) of AL-335 and Its Metabolite (ALS-022399 and ALS-022227)
Description: Clast is the last measurable plasma concentration (Clast) of AL-335, ALS-022399 and ALS-022227. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
ng/ml
  AL-335 | 5.931 (4.752) | 7.077 (4.676) | 4.983 (3.339) | 5.698 (5.620) | 5.811 (8.622)
  ALS-022399 | 5.995 (1.649) | 10.335 (5.558) | 14.591 (10.741) | 14.793 (8.738) | 17.520 (10.972)
  ALS-022227 | 38.28 (12.20) | 47.26 (10.68) | 67.08 (40.66) | 69.18 (38.01) | 72.14 (29.23)

19. Secondary Outcome: Time Corresponding to Last Measurable Plasma Concentration (Tlast) for AL-335 and Its Metabolites (ALS-022399 and ALS-022227)
Description: Tlast is the time corresponding to last measurable plasma concentration for AL-335, ALS-022399 and ALS-022227. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
Hours
  AL-335 | 6.000 [6.00 to 9.00] | 6.000 [6.00 to 9.00] | 6.000 [4.00 to 24.10] | 6.025 [6.0 to 9.00] | 8.670 [5.98 to 12.00]
  ALS-022399 | 12.000 [9.00 to 12.00] | 12.000 [12.00 to 12.00] | 12.000 [9.00 to 24.10] | 12.000 [12.00 to 12.00] | 12.000 [8.50 to 24.00]
  ALS-022227 | 24.00 [24.0 to 24.1] | 24.00 [23.7 to 24.1] | 24.00 [24.0 to 24.1] | 24.00 [24.0 to 24.2] | 23.90 [23.5 to 24.0]

20. Secondary Outcome: Average Plasma Concentration at Steady State (Css,Avg) of ALS-022227
Description: Css,avg is the average plasma concentration at steady state of ALS-022227. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
ng/ml | 121.49 (42.81) | 135.20 (41.16) | 218.88 (81.80) | 217.17 (83.26) | 227.37 (78.46)

21. Secondary Outcome: Cmin of Simeprevir
Description: Cmin is the minimum measured plasma concentration of simeprevir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 16 | 6 | 27
ng/ml | 379.75 (247.02) | 452.65 (641.99) | 517.00 (416.45) | 561.19 (424.71)

22. Secondary Outcome: Cmax of Simeprevir
Description: Cmax is the maximum measured plasma concentration of simeprevir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 16 | 6 | 27
ng/ml | 1927.7 (1205.3) | 1537.6 (1325.2) | 1769.3 (881.6) | 1925.1 (1034.0)

23. Secondary Outcome: Ctrough of Simeprevir
Description: Ctrough is the trough plasma concentration of Simeprevir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 16 | 6 | 27
ng/ml | 475.42 (317.63) | 570.64 (816.36) | 669.00 (442.50) | 636.88 (455.94)

24. Secondary Outcome: Tmax of Simeprevir
Description: Tmax is the Time to reach the maximum plasma concentration of simeprevir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 16 | 6 | 27
Hours | 6.000 [4.00 to 12.00] | 6.000 [4.00 to 9.00] | 6.000 [4.00 to 6.05] | 6.000 [3.00 to 8.50]

25. Secondary Outcome: AUC (0-last) of Simeprevir
Description: AUC (0-last) is the area under the plasma concentration-time curve from time 0 to last measurable plasma concentration of simeprevir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Cohort 1 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 16 | 6 | 27
ng*h/ml | 25018.2 (15248.7) | 23061.3 (24724.4) | 25266.7 (15523.4) | 27070.7 (15895.7)

26. Secondary Outcome: AUC (0-24) of Simeprevir
Description: AUC (0-24) is the area under the plasma concentration-time curve from time 0 to 24 hours of simeprevir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, and 24 hours postdose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Cohort 1 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 16 | 6 | 27
ng*h/ml | 25018.2 (15248.7) | 23061.3 (24724.4) | 25266.7 (15523.4) | 27070.7 (15895.7)

27. Secondary Outcome: Clast of Simeprevir
Description: Clast is the maximum measured plasma concentration of simeprevir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 16 | 6 | 27
ng/ml | 402.55 (244.20) | 481.76 (644.76) | 538.67 (456.21) | 602.60 (453.12)

28. Secondary Outcome: Tlast of Simeprevir
Description: Tlast is the time corresponding to last measurable plasma concentration of simeprevir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 16 | 6 | 27
Hours | 24.00 [24.0 to 24.1] | 24.00 [24.0 to 24.1] | 24.00 [24.0 to 24.2] | 23.90 [23.5 to 24.0]

29. Secondary Outcome: Average Plasma Concentration at Steady State (Css,Avg) of Simeprevir
Description: Css,avg is the average plasma concentration at steady state of simeprevir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 16 | 6 | 27
ng/ml | 1042.8 (634.3) | 960.5 (1030.7) | 1053.8 (647.8) | 1134.6 (666.6)

30. Secondary Outcome: Cmin of Odalasvir
Description: Cmin is the minimum observed plasma concentration of odalasvir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
ng/ml | 322.45 (139.21) | 97.21 (58.62) | 107.90 (49.46) | 102.73 (47.08) | 131.31 (62.31)

31. Secondary Outcome: Cmax of Odalasvir
Description: Cmax is the maximum observed plasma concentration of odalasvir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
ng/ml | 634.27 (257.29) | 363.36 (184.48) | 322.46 (167.29) | 232.85 (187.53) | 298.67 (133.99)

32. Secondary Outcome: Ctrough of Odalasvir
Description: Ctrough is the trough plasma concentration of odalasvir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
ng/ml | 335.18 (146.14) | 100.98 (61.90) | 112.44 (51.53) | 119.82 (58.87) | 141.56 (64.81)

33. Secondary Outcome: Tmax of Odalasvir
Description: Tmax is the time to reach the maximum plasma concentration of odalasvir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
Hours | 6.000 [4.00 to 12.00] | 6.000 [4.00 to 12.00] | 6.000 [3.00 to 9.00] | 4.500 [0.00 to 9.00] | 6.000 [3.98 to 9.00]

34. Secondary Outcome: AUC (0-last) of Odalasvir
Description: AUC(0-last) is the area under the plasma concentration-time curve from time 0 to last measurable plasma concentration of odalasvir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
ng*h/ml | 11805.5 (4902.6) | 8635.5 (4656.7) | 8648.1 (4161.1) | 7050.0 (4001.4) | 8422.2 (3617.8)

35. Secondary Outcome: AUC (0-24) for Odalasvir
Description: AUC(0-24) is the area under the plasma concentration-time curve from time zero to time 24 hours for odalasvir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, and 24 hours postdose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
ng*h/mL | 11805.5 (4902.6) | 5530.0 (2930.3) | 5393.8 (2695.4) | 4048.3 (2727.8) | 4924.1 (2122.9)

36. Secondary Outcome: Clast of Odalasvir
Description: Clast is the last measurable plasma concentration (Clast) of odalasvir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
ng/ml | 384.09 (172.29) | 162.65 (87.39) | 163.54 (78.10) | 131.92 (74.01) | 152.47 (66.50)

37. Secondary Outcome: Tlast of Odalasvir
Description: Tlast is the time corresponding to last measurable plasma concentration of odalasvir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
Hours | 24.00 [24.0 to 24.1] | 47.60 [47.5 to 47.7] | 47.50 [47.4 to 47.9] | 47.80 [47.4 to 48.0] | 47.50 [47.5 to 47.9]

38. Secondary Outcome: Average Plasma Concentration at Steady State (Css,Avg) of Odalasvir
Description: Css,avg is the average plasma concentration at steady state of odalasvir. For PK analyses, cohorts were grouped by treatment dosage (not duration of treatment) for participants without cirrhosis (Cohort 1; Cohort 1b+4; Cohort 2+3+5) and for participants with cirrhosis (Cohort 6; Cohort 7+8+9+11).
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 1b + Cohort 4 | Cohort 2 + Cohort 3 + Cohort 5 | Cohort 6 | Cohort 7 + Cohort 8 + Cohort 9 + Cohort 11
Number analyzed (Participants) | 11 | 11 | 16 | 6 | 27
ng/ml | 491.55 (203.85) | 181.60 (97.99) | 181.58 (87.25) | 147.40 (83.86) | 176.86 (75.91)

39. Secondary Outcome: Percentage of Participants With Virologic Relapse During the Follow-up Period
Description: Viral relapse is defined as participants SVR12, with HCV RNA <LLOQ at the actual end of study drug treatment and confirmed HCV RNA greater than or equal to (>=) LLOQ during follow up.
Time Frame: Follow up period (Up to Week 12 after end of treatment)
Population: Safety set included all participants enrolled into study who had received at least 1 dose of any study drug, whether prematurely withdrawn from study or not.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Percentage of participants | 0 | 16.0 | 0 | 0 | 0 | 100.0 | 14.3 | 3.3 | 0 | 0

40. Secondary Outcome: Percentage of Participants With On-treatment Failure
Description: On-treatment failure was defined by participants who did not achieve SVR12 and with confirmed HCV RNA >= LLOQ at the actual end of study drug treatment.
Time Frame: Up to 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Percentage of participants | 0 | 0 | 0 | 0 | 12.5 | 0 | 7.1 | 0 | 0 | 0

41. Secondary Outcome: Percentage of Participants Who Achieved HCV RNA Less Then (<) LLOQ Undetectable
Description: Percentage of participants who achieved HCV RNA less then (<) LLOQ undetectable was reported.
Time Frame: Day 2, 3, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 and End of treatment (Cohort 3: 6 weeks; Cohort 1, Cohort 1b+ Cohort 4, Cohort 2, Cohort 5a, and Cohort 6, 7, 8: 8 weeks; Cohort 4, Cohort 5b, Cohort 9 and Cohort 11: 12 weeks)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Percentage of participants
  Day 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 3 | 0 | 0 | 0 | 5.0 | 0 | 0 | 0 | 0 | 6.7 | 0
  Week 1 | 5.0 | 20.0 | 0 | 30.0 | 12.5 | 20.0 | 35.7 | 16.7 | 13.3 | 25.0
  Week 2 | 35.0 | 44.0 | 45.0 | 70.0 | 25.0 | 40.0 | 64.3 | 50.0 | 66.7 | 75.0
  Week 3 | 70.0 | 76.0 | 75.0 | 80.0 | 62.5 | 60.0 | 85.7 | 73.3 | 86.7 | 100
  Week 4 | 80.0 | 92.0 | 90.0 | 85.0 | 87.5 | 60.0 | 92.9 | 80.0 | 86.7 | 100
  Week 5 | 100 | 96.0 | 100 | 90.0 | 100 | 80.0 | 92.9 | 90.0 | 100 | 100
  Week 6 | 90.0 | 100 | 85.0 | 90.0 | 100 | 100 | 92.9 | 96.7 | 100 | 100
  Week 7 | 90.0 | 96.0 | 95.0 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 6. | 100 | 80.0 | 85.7 | 100 | 100 | 100
  Week 8 | 95.0 | 100 | 100 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 6. | 87.5 | 100 | 85.7 | 100 | 93.3 | 100
  Week 9 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 6. | 87.5 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 92.9 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 93.3 | 100
  Week 10 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 6. | 87.5 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 92.9 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 93.3 | 100
  Week 11 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 6. | 87.5 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 92.9 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 86.7 | 100
  Week 12 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 6. | 87.5 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 85.7 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 93.3 | 100
  End of treatment | 95.0 | 100 | 100 | 90.0 | 87.5 | 100 | 85.7 | 100 | 93.3 | 100

42. Secondary Outcome: Percentage of Participants Who Achieved HCV RNA <LLOQ
Description: Percentage of participants who achieved HCV RNA <LLOQ was reported.
Time Frame: as for outcome 41
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 20 | 25 | 20 | 20 | 8 | 5 | 14 | 30 | 15 | 4
Percentage of participants
  Day 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 1 | 0 | 8.0 | 0 | 10.0 | 0 | 0 | 14.3 | 16.7 | 13.3 | 25.0
  Week 2 | 20.0 | 20.0 | 15.0 | 40.0 | 0 | 20.0 | 42.9 | 50.0 | 66.7 | 75.0
  Week 3 | 40.0 | 40.0 | 45.0 | 65.0 | 37.5 | 60.0 | 50.0 | 73.3 | 86.7 | 100
  Week 4 | 55.0 | 52.0 | 60.0 | 80.0 | 62.5 | 40.0 | 78.6 | 80.0 | 86.7 | 100
  Week 5 | 75.0 | 96.0 | 85.0 | 85.0 | 75.0 | 80.0 | 85.7 | 90.0 | 100 | 100
  Week 6 | 80.0 | 88.0 | 85.0 | 80.0 | 87.5 | 80.0 | 92.9 | 96.7 | 100 | 100
  Week 7 | 80.0 | 92.0 | 95.0 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 6. | 87.5 | 80.0 | 85.7 | 100 | 100 | 100
  Week 8 | 85.0 | 96.0 | 100 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 6. | 87.5 | 100 | 85.7 | 100 | 93.3 | 100
  Week 9 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 6. | 87.5 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 92.9 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 93.3 | 100
  Week 10 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 6. | 87.5 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 92.9 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 93.3 | 100
  Week 11 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 6. | 87.5 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 92.9 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 86.7 | 100
  Week 12 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | NA — NA indicates that the data was not estimable for the specified timepoint. | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 6. | 87.5 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 78.6 | NA — NA indicates that data was not collected at this timepoint since participants in this arm ended treatment at week 8. | 93.3 | 100
  End of treatment | 85.0 | 96.0 | 100 | 80.0 | 87.5 | 100 | 78.6 | 100 | 93.3 | 100

43. Secondary Outcome: Time to Achieve Undetectable HCV RNA or < LLOQ HCV RNA
Description: Time to achieve undetectable HCV RNA or < LLOQ HCV RNA was reported.
Time Frame: Up to Week 24 (follow up visit)
Population: Safety set included all participants enrolled into the study who had received at least 1 dose of any study drug, whether prematurely withdrawn from the study or not. Data was not collected and analyzed for this outcome measure as per the change in planned analysis.
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

44. Secondary Outcome: Number of Participants With HCV Nonstructural Protein NS5A, NS5B, and NS3/4A Sequence in Participants With Virologic Failure
Description: Sequencing of the HCV nonstructural protein 3/4A (NS3/4A), nonstructural protein 5A (NS5A) and nonstructural protein 5B (NS5B) genes was done to identify pre-existing sequence polymorphisms and characterize emerging HCV viral variants in participants with virologic failure.
Time Frame: Up to Week 24 (Follow up visit)
Population: Safety set included all participants enrolled into the study who had received at least 1 dose of any study drug, whether prematurely withdrawn from the study or not. Participants who had virologic failure were included in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
Number analyzed (Participants) | 0 | 4 | 0 | 0 | 1 | 5 | 3 | 1 | 0 | 0
Participants |  | 4 |  |  | 1 | 0 | 2 | 1 |  |

ADVERSE EVENTS:
Time Frame: Up to 43 weeks
Description: Safety set included all participants enrolled into the study who had received at least 1 dose of any study drug, whether prematurely withdrawn from the study or not.
Arm/Group | Cohort 1 (8 Weeks Genotype [GT1]) | Cohort 1b + Cohort 4 (8 Weeks GT1) | Cohort 2 (8 Weeks GT1) | Cohort 3 (6 Weeks GT1) | Cohort 4 (12 Weeks GT1) | Cohort 5a (8 Weeks GT3) | Cohort 5b (12 Weeks GT3) | Cohort 6,7,8 (8 Weeks GT1 F4) | Cohort 9 (12 Weeks GT1 F4) | Cohort 11 (12 Weeks GT2 F4)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/25 | 0/20 | 0/20 | 0/8 | 0/5 | 0/14 | 0/30 | 0/15 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/20 | 2/25 | 0/20 | 0/20 | 0/8 | 0/5 | 0/14 | 1/30 | 2/15 | 1/4
Other Adverse Events (participants affected / at risk) | 17/20 | 20/25 | 14/20 | 14/20 | 7/8 | 4/5 | 13/14 | 18/30 | 10/15 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (8 Weeks Genotype [GT1]) (N=20) | Cohort 1b + Cohort 4 (8 Weeks GT1) (N=25) | Cohort 2 (8 Weeks GT1) (N=20) | Cohort 3 (6 Weeks GT1) (N=20) | Cohort 4 (12 Weeks GT1) (N=8) | Cohort 5a (8 Weeks GT3) (N=5) | Cohort 5b (12 Weeks GT3) (N=14) | Cohort 6,7,8 (8 Weeks GT1 F4) (N=30) | Cohort 9 (12 Weeks GT1 F4) (N=15) | Cohort 11 (12 Weeks GT2 F4) (N=4)
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transitional Cell Carcinoma Urethra (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (8 Weeks Genotype [GT1]) (N=20) | Cohort 1b + Cohort 4 (8 Weeks GT1) (N=25) | Cohort 2 (8 Weeks GT1) (N=20) | Cohort 3 (6 Weeks GT1) (N=20) | Cohort 4 (12 Weeks GT1) (N=8) | Cohort 5a (8 Weeks GT3) (N=5) | Cohort 5b (12 Weeks GT3) (N=14) | Cohort 6,7,8 (8 Weeks GT1 F4) (N=30) | Cohort 9 (12 Weeks GT1 F4) (N=15) | Cohort 11 (12 Weeks GT2 F4) (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Porphyria Non-Acute (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear Discomfort (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear Pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry Eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema of Eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye Pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual Impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Loose Tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Noninfective Sialoadenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Salivary Gland Calculus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Chest Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Chest Pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 4 | 2 | 3 | 2 | 0 | 6 | 3 | 1 | 2
Feeling Abnormal (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel Puncture Site Bruise (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Vessel Puncture Site Haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vessel Puncture Site Phlebitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angular Cheilitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash Pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 3 | 1 | 1 | 3 | 2 | 4 | 3 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Chest Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 4 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lip Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Creatine Phosphokinase Increase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ejection Fraction Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram Pr Prolongation (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appetite Disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyperphagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 3 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Burning Sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disturbance in Attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 8 | 5 | 2 | 3 | 4 | 2 | 3 | 2 | 2 | 1
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyposmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Memory Impairment (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sensory Disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tension Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal Dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depressed Mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flat Affect (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Libido Decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Panic Attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hand Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mechanical Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Limitations of the study included the open-label design, limited sample size, and the lack of a comparator group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT02569710/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT02569710/SAP_001.pdf